CLINICAL TRIAL: NCT06936280
Title: A Group-based Psychological Intervention for Emerging Adults With Type 1 Diabetes and Diabetes Distress
Brief Title: Type 1 Diabetes and Diabetes Distress
Acronym: ACTnow
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Steno Diabetes Center Odense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25/13117; 25/13117 (Other: Steno Diabetes Center Odense)
Record Dates: First submitted 2025-03-31; First posted 2025-04-20 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Distress; Diabetes Mellitus Type 1
Keywords: RCT study; type 1 diabetes; diabetes distress; ACTnow
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Waiting list design. Randomization to either a control group or intervention group. The intervention group will receive the intervention at T0 whereas the control group will wait 3 months before receiving the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention at t0 (Experimental)
  Interventions: Behavioral: ACTnow
- wait list control group (Experimental): Control group for the first 3 months, whereafter the arm will receive the same intervention as arm 1
  Interventions: Behavioral: ACTnow

INTERVENTIONS:
Behavioral: ACTnow — The group-based psychological intervention consists of six bi-weekly sessions, each lasting two hours, with 6-10 participants per group, led by a psychologist and nurse.
  The intervention is based on Acceptance and Commitment Therapy (ACT), an evidence-based approach shown to be effective for chronic diseases, with additional elements from cognitive behavioral therapy and health education. It is manual-based, developed by experienced clinicians at SDCO, and includes tools from an existing diabetes distress intervention (REDUCE).
  Each session includes a mindfulness exercise, a review of the previous session, a new topic, individual homework assignments, and a conclusion. Participants complete an online questionnaire to track diabetes distress after each session. The group process lasts about 3 months. Preliminary results from a feasibility study showed positive outcomes in recruitment, patient satisfaction, and reduction of diabetes distress (publication in progress).

SUMMARY:
The goal of this clinical trial is to reduce diabetes distress in emerging adults (18-35 years) with type 1 diabetes and moderate-to-severe diabetes distress.

The expectation is that a group-based psychological intervention (ACTnow) will not only reduce diabetes distress but also improve psychological well-being and glycemic outcomes.

The intervention involves a multidisciplinary team, including nurses, psychologists, and physicians, and is designed in a format that can easily be integrated into future standard care.

The main research questions are:

* Does a group-based psychological intervention reduce diabetes distress?
* Does a group-based psychological intervention improve psychological well-being and glycemic outcomes?

Researchers will compare the group-based psychological intervention (arm 1) with a waitlist control group, which will receive the intervention after three months (arm 2).

Participants will first attend a virtual screening interview with a psychologist or nurse to identify if they are eligible to participate in the study. After randomization, the intervention group receives six bi-weekly sessions, each lasting two hours, led by a psychologist and nurse. Each session includes a mindfulness exercise, a review of the previous session, a new topic, individual homework assignments, and a conclusion.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 6 months
* Age between 18 and 35
* T1-DDS score ≥ 2, or T1-DDS subscale score ≥ 2
* Treated in a diabetes clinic in the Region of Southern Denmark
* Proficient in Danish

Exclusion Criteria:

* Psychiatric diagnosis: diagnosed with substance abuse, alcohol abuse, psychosis, schizophrenia or any other psychiatric diagnosis that may compromise participation in the intervention
* Cognitive disorders such as brain injury
* Complex challenges best suited to individual treatment
* Current therapeutic treatment for depression, anxiety or stress
* Not stable medication for anxiety/depression for the past two months or planned change in medication for anxiety/depression during the project period

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in diabetes distress score using T1-DDS | from baseline to 3 months
  The primary outcome, is a reduction in the degree of diabetes distress measured using the Type 1 Diabetes Distress Scale (T1-DDS). The scale uses a 6 point likert-scale. The combined DDS score is divided by 28 to give a number between 1 and 6. A score between 2,00-2,99 is defined as moderate diabetes distress, and a score above 3,00 is defined as high diabetes distress.

SECONDARY OUTCOMES:
Change in the T1-DDAS score | from baseline to 3 months
  Using the Type 1-Diabetes Distress Assessment System to assess change in concerns related to diabetes technology. 5 point likert scale. A score above 2,00 is consideret moderat concerns.
Change in AADQ score | from baseline to 3 months
  Using The Acceptance and Action Diabetes Questionnaire (AADQ) to assess change in acceptance of thoughts and feelings about diabetes. 7 point likert scale.
Change in GAD-7 score | from baseline to 3 months
  Using the Generalized Anxiety Disorder Assessment (GAD-7) to assess change in symptoms of anxiety. Using a 4 point likert scale. A score between 15-21 is consideret great anxiety.
Change in HbA1c | from baseline to 3 months
  Improved blood glucose control measured by HbA1c. Either reduced or increased HbA1c, depending on the patient
Change in PHQ-9 score | from baseline to 3 months
  Reduced symptoms of depression using the Patient Health Questionnaire (PHQ-9). 4 point likert scale. a score of 20-27 is considered great depression

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Esbjerg Hospital, Esbjerg
  - Odense University Hospital, Odense
  - Sønderborg Hospital, Sønderborg

IPD SHARING:
Plan to Share IPD: No